CLINICAL TRIAL: NCT07280338
Title: Emotional Intelligence and Chronic Orofacial Pain
Acronym: IEDOF
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0372; 2025-A00682-47 (Registry Identifier: ANSM - IDRCB)
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pain
Keywords: Emotional intelligence
MeSH Terms: conditions — Chronic Pain | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Evaluation of the potential link between emotional intelligence and chronic orofacial pain.: All included subjects will have the same participation, which consists of completing several standardized questionnaires. These questionnaires assess various psychological and emotional aspects, including anxiety and depressive disorders (HADS questionnaire), coping strategies (Brief-COPE score), emotional regulation (ERS score), fatigue level (EVA scale), and emotional intelligence (TEIQue-SF questionnaire) to compare scores between the DTM group and the control group. Additionally, sociodemographic and psychosocial criteria will be collected to refine the analysis of the results. The completion of these questionnaires is part of routine consultations and does not alter the patients' standard care.
  Interventions: Other: Questionnaire and Physical Exam

INTERVENTIONS:
Other: Questionnaire and Physical Exam — All included subjects will be required to complete the following questionnaires:
  Hospital Anxiety and Depression Scale (HADS) Brief-COPE for coping assessment Emotion Reactivity Scale (ERS) for emotional regulation Visual Analog Scale (VAS) for fatigue assessment Sociodemographic and psychosocial evaluation Trait Emotional Intelligence Questionnaire - Short Form (TEIQue-SF) for emotional intelligence assessment

SUMMARY:
Chronic pain, lasting more than three months, is a widespread health issue that negatively impacts daily life, leading to significant emotional distress and functional impairment. Emotional intelligence, defined as the ability to recognize and manage one's own emotions as well as those of others, has been linked to better communication skills and reduced stress, which is a well-known risk factor for chronic pain. Studies have highlighted a correlation between emotional intelligence and certain chronic pain conditions, such as fibromyalgia and migraines. However, no research has yet explored its role in painful temporomandibular disorders (TMD). Given the strong involvement of psychosocial factors in TMD etiology, a better understanding of these elements could improve pain management and pave the way for preventive interventions.

DETAILED DESCRIPTION:
This project aims to compare emotional intelligence and various psychosocial factors (anxiety, depression, coping, emotional regulation) between patients with painful temporomandibular disorder (TMD) and a control group without TMD or chronic pain. The study is based on the administration of validated French-language questionnaires during routine dental medicine consultations. Each participant completes these questionnaires in approximately 15 minutes, without any modification to their care. The data collected will help assess the relationships between orofacial pain and emotional factors to improve the understanding and management of affected patients.

ELIGIBILITY:
Inclusion Criteria:

For all subjects:

Major subject

* Non-opposition obtained
* For subjects in the TMD group:

Diagnosis of temporomandibular dysfunction -No other diagnosis of chronic pain

For subjects in the control group:

-No diagnosis of chronic pain

Non inclusion Criteria:

* Subject not understanding French
* Subject under legal protection (guardianship or curatorship)
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Regarding the evaluated population (cases), approximately 30 patients are seen each week in the oral health service for chronic orofacial pain consultations. About 60% of these patients have a diagnosis of painful TMD, which is around 18 patients per week. Including 44 patients in this study over a 6-month period thus seems feasible.
  Regarding the control population, more than 50 patients are seen daily in oral rehabilitation consultations at the oral health service of the CHU de Brest. These controls will be matched in gender and age (+/- 5 years) with the studied population (cases). The significant proportion of these patients should allow for the feasibility of this matching.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of emotional intelligence score between both groups | Day 0
  Measurement of emotional intelligence score assessed by the TEIQue-SF questionnaire :
  The short version consists of 33 items assessing four factors: well-being, self-control, emotionality, and sociability. Each item is rated on a Likert scale ranging from 1 ("strongly disagree") to 7 ("strongly agree").

SECONDARY OUTCOMES:
Measurement of anxiety disorders between both groups | Day 0
  Measurement of anxiety disorders between the two groups via the HAD-S questionnaire
  The HAD scale is a validated instrument in French, used to screen for anxiety and depressive disorders. It consists of 14 items scored from 0 to 3. Seven questions relate to anxiety (total A) and the other seven to the depressive dimension (total D), thus providing two scores (maximum score for each = 21). This questionnaire is routinely used during consultations in the oral health service and systematically used during specialized consultations for orofacial pain.
Measurement of the coping score between both groups | Day 0
  Measurement of the coping score assessed by the Brief-COPE questionnaire
  This instrument is an abbreviated version of the COPE inventory with 28 items. It includes 14 scales that assess distinct dimensions of coping: active coping, planning, instrumental social support seeking, emotional social support seeking, emotional expression, behavioral disengagement, distraction, blaming, positive reinterpretation, humor, denial, acceptance, religion, and substance use.
Measurement of emotional regulation score between both groups | Day 0
  Measurement of emotional regulation score assessed by the ERS questionnaire
  The ERS is a self-report questionnaire with 21 items designed to measure, using a single tool, three dimensions of emotional reactivity: emotional sensitivity, intensity, and persistence of emotions. Each item is rated on a Likert scale ranging from 0 ("does not apply to me at all") to 4 ("applies to me perfectly").
Measurement of fatigue score between both groups | Day 0
  Measurement of fatigue score assessed by an EVA scale (From 0 to 10)
Measurement of Depression disorders between both groups | Day 0
  Measurement of depression disorders between both groups via the HAD-S questionnaire
  The HAD scale is a validated instrument in French, used to screen for anxiety and depressive disorders. It consists of 14 items scored from 0 to 3. Seven questions relate to anxiety (total A) and the other seven to the depressive dimension (total D), thus providing two scores (maximum score for each = 21). This questionnaire is routinely used during consultations in the oral health service and systematically used during specialized consultations for orofacial pain.

IPD SHARING:
Plan to Share IPD: Undecided